CLINICAL TRIAL: NCT01905501
Title: Sevoflurane Protective Effect on Ischemia-reperfusion Injury in Patients Undergoing Reconstructive Plastic Surgery With Microsurgical Flap. Multicenter, Randomized Controlled Trial.
Brief Title: Sevoflurane Protective Effect on Ischemia-reperfusion Injury. Multicenter, Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Ester Forastiere, M.D., Chief of Critical Area Department, Regina Elena Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Versione 02.01.2013
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Microsurgical Free Flaps
Keywords: Balanced anesthesia; Inhalation anesthesia; Reperfusion injury; Microsurgical Free flap
MeSH Terms: conditions — Reperfusion Injury | interventions — Balanced Anesthesia; Anesthesia, Inhalation

ARMS (2):
- Total intravenous anesthesia (Active Comparator): Total intravenous anaesthesia
  Interventions: Drug: Total intravenous anesthesia
- Balanced anesthesia (Experimental)
  Interventions: Drug: Balanced anesthesia

INTERVENTIONS:
Drug: Balanced anesthesia — Et-Sevo maIntained 1,8-2%, remifentanyl according target-controlled infusion maintained 1-3 ng/ml
  Other Names: Inhalation anesthesia
  Arms: Balanced anesthesia
Drug: Total intravenous anesthesia — Propofol 3-4 µg/ml and remifentanyl 1-3 ng/ml according target-controlled infusion
  Other Names: TIVA-TCI
  Arms: Total intravenous anesthesia

SUMMARY:
This study aimed to evaluate the possible protective effect of anesthetic technique balanced(with sevoflurane) compared with total intravenous anesthetic technique (propofol,remifentanil). The hypothesis is that the Sevoflurane may exert protective effect in regard to the ischemia-reperfusion injury induced on the microsurgical breast free flap during transfer to receiving area. The investigators will evaluate the continuous flap tissue oximetry and the level of biochemical markers.

ELIGIBILITY:
Inclusion Criteria:

Patient selected for plastic breast surgery With microsurgical Free flap Over 18 y Asa I/II

Exclusion Criteria:

Unusual reaction to anesthetic drugs Suspect for malignant hyperthermia Vasculopathic disease Coagulation disease

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
continuous tissue oximetry (NIRS) | 20 hours

SECONDARY OUTCOMES:
Biochemical Markers | Preoperative and 24 hours post operative
Lactate Clearance | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ester Forastiere, M.D., Principal Investigator — Regina Elena CI
Locations (1):
- Regina Elena CI, Rome, Italy, Italy

REFERENCES:
- [Derived] Claroni C, Torregiani G, Covotta M, Sofra M, Scotto Di Uccio A, Marcelli ME, Naccarato A, Forastiere E. Protective effect of sevoflurane preconditioning on ischemia-reperfusion injury in patients undergoing reconstructive plastic surgery with microsurgical flap, a randomized controlled trial. BMC Anesthesiol. 2016 Aug 22;16(1):66. doi: 10.1186/s12871-016-0230-1. PMID 27549313